CLINICAL TRIAL: NCT02453360
Title: Impact of Volume of Local Anesthetic Injected for Adductor Canal Block on Recovery Profile and Block Characteristics Following Total Knee Arthroplasty.
Brief Title: Adductor Canal Block for Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2014-1419
Record Dates: First submitted 2015-05-11; First posted 2015-05-25 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Arthroplasty, Replacement, Knee; Pain, Postoperative
Keywords: Anesthesia; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 5 ml (Experimental): Following negative aspiration, SSACNB volume will be randomized and subjects will receive 5, 10 or 20 ml of 0.5% bupivacaine will be incrementally injected. Randomization of the volume of bupivacaine will be determined by opening a sequential, pre-sealed envelope with the group assignment designated within. All studied volumes are well within the acceptable range for SSACNB.
  Interventions: Procedure: Adductor Canal Block; Drug: Adductor Canal Block
- 10 ml (Experimental): Following negative aspiration, SSACNB volume will be randomized and subjects will receive 5, 10 or 20 ml of 0.5% bupivacaine will be incrementally injected. Randomization of the volume of bupivacaine will be determined by opening a sequential, pre-sealed envelope with the group assignment designated within. All studied volumes are well within the acceptable range for SSACNB.
  Interventions: Procedure: Adductor Canal Block; Drug: Adductor Canal Block
- 20 ml (Experimental): Following negative aspiration, SSACNB volume will be randomized and subjects will receive 5, 10 or 20 ml of 0.5% bupivacaine will be incrementally injected. Randomization of the volume of bupivacaine will be determined by opening a sequential, pre-sealed envelope with the group assignment designated within. All studied volumes are well within the acceptable range for SSACNB.
  Interventions: Procedure: Adductor Canal Block; Drug: Adductor Canal Block

INTERVENTIONS:
Procedure: Adductor Canal Block — Following negative aspiration, SSACNB volume will be randomized and subjects will receive 5, 10 or 20 ml of 0.5% bupivacaine will be incrementally injected. Randomization of the volume of bupivacaine will be determined by opening a sequential, pre-sealed envelope with the group assignment designated within. All studied volumes are well within the acceptable range for SSACNB.
Drug: Adductor Canal Block — Following negative aspiration, SSACNB volume will be randomized and subjects will receive 5, 10 or 20 ml of 0.5% bupivacaine will be incrementally injected. Randomization of the volume of bupivacaine will be determined by opening a sequential, pre-sealed envelope with the group assignment designated within. All studied volumes are well within the acceptable range for SSACNB.
  Other Names: Bupivacaine

SUMMARY:
Total knee arthroplasty (TKA) can be associated with a large amount of postoperative pain. This pain can oftentimes be severe enough to limit participation in physical therapy and ultimately delay discharge resulting in increased cost. Several strategies have been developed in an effort to decrease postoperative pain following TKA while maintaining lower extremity strength and maximizing participation in physical therapy. Recently, adductor canal blockade has gained popularity as it is reported to provide analgesia to the anterior knee without resulting in significant quadriceps muscle weakness. However, few studies have carefully evaluated the impact of volume of injection of local anesthetic into the adductor canal on motor weakness or pain control. The ability to achieve similar pain control with decreased volumes of local anesthetic would allow the surgery team to apply more local anesthetic to posterior knee structures. Decreased volumes of local anesthetic may also be associated with a decreased risk of local anesthetic toxicity. This study aims to carefully evaluate this relationship using a physical therapy evaluation method that relies on both motor strength and pain control. In addition, the investigators hope to carefully evaluate motor strength using a novel method of strength measurement in an effort to further evaluate the impact of volume of injection of local anesthetic into the adductor canal on motor strength.

DETAILED DESCRIPTION:
Postoperative analgesia for total knee arthroplasty (TKA) is incredibly important as it allows for effective physical therapy and ultimately ensures proper function of the implanted joint hardware. Unfortunately, TKA is oftentimes associated with pain severe enough to limit participation in physical therapy which can ultimately result in prolonged hospitalizations and perhaps decreased joint function. A number of strategies have been reported to decrease the pain associated with TKA. Opioids are commonly utilized but they can be associated with a number of potential side effects including nausea, itching, respiratory depression, tolerance and the potential for abuse. Epidural analgesia has been utilized for postoperative analgesia but this strategy requires urinary catheterization (potential source of increased incidence of urinary tract infections), causes significant vasodilation with resulting hypotension and can cause bilateral lower extremity weakness that can undermine efforts at early physical therapy and rehabilitation. Femoral nerve blockade and femoral nerve catheters have the potential to decrease pain in the anterior knee but use of this technique is limited by incomplete analgesia and quadriceps motor weakness. Some groups have advocated for the substitution or addition of sciatic or obturator nerve blocks to femoral nerve blockade but this is at the expense of increased lower extremity weakness and little potential clinical benefit.1-5

In an effort to balance the need for effective postoperative analgesia with the need to maintain lower extremity muscle strength for active participation in physical therapy, a number of groups have begun to evaluate the adductor canal block. The adductor canal is located in the middle 1/3 of the thigh and includes the saphenous nerve and nerve to the vastus medialis. The primary advantage to adductor canal blockade versus femoral nerve blockade is a potential sparing of the nerves to the quadriceps muscle and therefore preservation of lower extremity motor strength.6-8 Kwofie et al reported in a study of 16 volunteers that there was no change in quadriceps strength or hip adduction following the injection of 15 ml of local anesthetic. This is interesting as the obturator nerve is reported to travel within the adductor canal and is responsible for hip adduction. Kwofie et al also reported that SSACNB resulted in significantly decreased impairments with balance compared to a SSFNB.9

To this point, the majority of studies evaluating adductor canal blockade have focused on continuous techniques and little has been done to evaluate single shot techniques. Continuous techniques have the potential to extend analgesia but this is at the expense of increased cost, effort, resource utilization and potentially increased risk of infection.

The safety of CACNB technique was highlighted by a study by Henningsen et al where no cases of nerve injury related to analgesic technique were reported in a series of 97 patients.10 Andersen et al compared a CACNB vs control in 40 patients and found that the intervention group reported decreased pain and sleep disturbances while retaining the ability to ambulate soon after surgery.11 Mudumbai et al evaluated 180 patients undergoing TKA and discovered that continuous adductor canal nerve blockade (CACNB) relative to continuous femoral nerve blockade (CFNB) resulted in greater ability to ambulate (37 m vs 6 m) on POD 1 and similar pain scores.8 Jaeger et al examined a similar group of 54 patients presenting for TKA and found that CACNB relative to CFNB resulted in decreased quadriceps weakness and no difference in pain, opioid consumption or weakness.12 Jenstrup et al reported that, compared to placebo, CACNB resulted in decreased pain with flexion and opioid consumption.13 Only recently has a study comparing SSACNB and SSFNB been published. This study demonstrated that SSACNB resulted in decreased postoperative quadriceps weakness and similar pain control to SSFNB.14 Of interest, previous research has demonstrated that 15 ml 0.5% ropivacaine is required to produce ultrasound guided femoral nerve blockade (including sensory and quadriceps motor weakness) but no such study has yet been done for the adductor canal block.15 It is possible that larger volumes of local anesthetic injected into the adductor canal could result in proximal spread of local anesthetic and increase quadriceps weakness and difficulty ambulating. It is also possible that decreased volumes of injection may result in inferior pain control and difficulties participating in physical therapy.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is scheduled for elective unilateral TKA
2. The subject is ≥ 18 years and ≤ 80 years;
3. The subject's weight is between 70-120 kg; and
4. The subject's primary anesthesia care team has planned for a neuraxial anesthetic (i.e. spinal, epidural or combined-spinal epidural).
5. The patient agrees to receive an adductor canal block.
6. American Society of Anesthesiologists class 1-3

Exclusion Criteria:

1. Subject is < 18 years of age or >80 years of age;
2. Subject is non-English speaking;
3. Subject is known or believed to be pregnant;
4. Subject is a prisoner;
5. Subject has impaired decision-making capacity; per discretion of the Investigator
6. Symptomatic untreated gastroesophageal reflux or otherwise at risk for perioperative aspiration;
7. Any condition for which the primary anesthesia care team deems neuraxial anesthesia inappropriate;
8. Significant pre-existing neuropathy on the operative limb;
9. Significant renal, cardiac or hepatic disease per discretion of the investigator.
10. American Society of Anesthesiologists class 4-5
11. Known hypersensitivity and/or allergies to local anesthetics
12. Chronic Opioid Use (daily or almost daily use of opioids for > 3 months)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-05; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5 ml | 10 ml | 20 ml
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 ml | 10 ml | 20 ml | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (6.9) | 62.6 (7.8) | 62 (7.6) | 63.1 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 14 | 39
  Male | 10 | 5 | 6 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60
Body Mass Index kg/m2 [Mean (Standard Deviation); unit: kg/m^2] | 31.1 (3.8) | 34.3 (6) | 34.2 (5.9) | 33.2 (5.5)
ASA Physical Status Classification System Score [Median (Full Range); unit: units on a scale] — Measure Description: ASA I- A normal healthy patient. ASA II- A patient with mild systemic disease. ASA III- A patient with severe systemic disease. ASA IV- A patient with severe systemic disease that is a constant threat to life.
  ASA V- A moribund patient who is not expected to survive without the operation. ASA VI- A declared brain-dead patient whose organs are being removed for donor purposes.
  units on a scale | 2 [1 to 3] | 2 [1 to 2] | 2 [2 to 3] | 2 [1 to 3]

OUTCOME MEASURES:

1. Primary Outcome: 10 Meter Walk Test
Description: This will be evaluated by determining how quickly a patient is able to ambulate over 10 meters on POD 1 (10 meter walk test).
Time Frame: 24 hours postoperatively following total knee arthroplasty
Population: Incomplete data responsible for discrepancies between number of subjects enrolled and data reported.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | 5 ml | 10 ml | 20 ml
Number analyzed (Participants) | 19 | 18 | 16
Seconds | 38.6 (33.3) | 49.8 (55.4) | 43.3 (31.5)

2. Secondary Outcome: Opioid Consumption
Description: Opioid Requirements will be retrieved from the patient's electronic medical record
Time Frame: PACU Discharge through 24 hours postoperatively
Measure: Mean (Standard Deviation); unit: Morphine Equivalents (mg)
Arm/Group | 5 ml | 10 ml | 20 ml
Number analyzed (Participants) | 20 | 20 | 20
Morphine Equivalents (mg) | 33.8 (20.5) | 30.9 (16.2) | 29.1 (14.6)

3. Secondary Outcome: Pain With Activity at 24 Hours
Description: Patient pain will be assessed by having participants describe pain using Numerical Ranking Scale (NRS) with a total score of 0-10 where 0 is no pain and 10 is the worst pain imaginable. Location of pain will also be assessed.
Time Frame: 24 Hours Following Surgery
Population: Incomplete data responsible for discrepancies between number of subjects enrolled and data reported.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 5 ml | 10 ml | 20 ml
Number analyzed (Participants) | 19 | 19 | 20
Scores on a scale | 5 (2) | 5 (2) | 6 (1.9)

4. Secondary Outcome: Percentage Change in Knee Extension Strength From Baseline
Description: Patient strength will be assessed by asking subjects to maximally adduct their leg or extend their knee for five seconds. Subjects will be asked to repeat this measurement three times at each measurement (pre-block, 15 minutes post-block, 24 hours post-block and 48 hours post-block). Strength measurements will be made with the Kiio strength monitoring device.
Time Frame: 24 Hours Following Surgery
Population: Incomplete data responsible for discrepancies between number of subjects enrolled and data reported.
Measure: Mean (Standard Deviation); unit: percentage change of Baseline Strength
Arm/Group | 5 ml | 10 ml | 20 ml
Number analyzed (Participants) | 17 | 18 | 17
percentage change of Baseline Strength | -59.7 (28.1) | -55 (24) | -64.3 (21.4)

5. Secondary Outcome: Number of Participants With Nausea at 24 Hours
Description: Need for antiemetic therapy will be assessed through evaluation of the electronic medical record.
Time Frame: Perioperative through 48 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | 5 ml | 10 ml | 20 ml
Number analyzed (Participants) | 20 | 20 | 20
Participants | 11 | 11 | 6

ADVERSE EVENTS:
Time Frame: 48 Hours
Arm/Group | 5 ml | 10 ml | 20 ml
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT02453360/Prot_SAP_000.pdf